CLINICAL TRIAL: NCT07394894
Title: Local Percutaneous Pulsed Radiofrequency Ablation Versus Ultrasound Guided Steroids Injection in Management of Pain in Cases of Chronic Planter Fascitis, Randomised Double Blinded Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Gamal Khafagy, Resident doctor at Anesthesia, Intensive Care and Pain Management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPC RA VS US steroids
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Planter Fascitis
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Local percutaneous pulsed radiofrequency Ablation PRFA was applied at 42 °C for eight minutes at 20 m/s intervals, aiming for an impedance of 250-500 ohms
  Interventions: Procedure: Local percutaneous pulsed radiofrequency Ablation PRFA
- Group B (Active Comparator): locally injection of steroids under ultrasound guided in planter fascitis ( 1ml containing 40 mg methylprednisolone)
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Procedure: Local percutaneous pulsed radiofrequency Ablation PRFA — Local percutaneous pulsed radiofrequency Ablation PRFA was applied at 42 °C for eight minutes at 20 m/s intervals, aiming for an impedance of 250-500 ohms
  Arms: Group A
Drug: methylprednisolone — locally injection of steroids under ultrasound guided in planter fascitis ( 1ml containing 40 mg methylprednisolone)
  Arms: Group B

SUMMARY:
Plantar fasciitis is the one of the most common causes of painful heel in adults. It is assumed to be caused by inflammation and is typically precipitated by biomechanical stress. It is very difficult to treat this condition as the causation is not exactly diagnosed (1) Plantar fascia is a broad band of fibrous tissue which originates from the anteromedial plantar aspect of the calcaneal tuberosity and inserts through several slips into the plantar aspects of the metatarsophalangeal joints, the flexor tendon sheaths, and the bases of the proximal phalanges of the digits. Athletic population has a high frequency of plantar fasciitis and in the non-athletic population it is most frequently seen in weight bearing occupations (2) Excessive pulling and stretching of plantar fascia either from excessive exercise or overuse, repeated trauma, aging, obesity, poor fitting shoe gear or poor foot alignment while running or prolong standing, produce microscopic tear of collagen or cystic degeneration in the origin of plantar fascia causing pain and inflammation.(3) Planter Fasciitis is considered a self limited condition. However, the long interval is frustrating for both patients and clinicians. Although, there are numerous reports describing operative and non-operative treatment options that claim to hasten the resolution of symptoms, few entail high level evidence to substantiate their claims. Without high quality data to identify which treatments are successful, the clinical decision making in the management of this condition is at times arbitrary and anecdotal (4) 3 The classic presentation of plantar fasciitis is pain on the sole of foot at the inferior region of the heel which is particularly worse with the first step taken after bed (5) Noninvasive Treatments PF is usually a self-limiting condition, with more than 90% of patients achieving symptomatic relief with 3-6 months of conservative treatment. 39 Initial treatment should consist of nonsteroidal antiinflammatories (NSAIDs), stretching of the gastrocnemius and the plantar fascia, and the use of an orthosis (heel pads, heel cups, arch supports, or night splints). Successful treatment is defined as a decrease in pain and improvement in function. Minimally Invasive Treatments Patients with heel pain for 6 months or more that is recalcitrant to the nonoperative treatments may undergo minimally invasive procedures that relieve pain (corticosteroid injection), decrease heel cord tightness (botulinum toxin injection), or stimulate the body's healing response (platelet rich plasma [PRP] injection, dry needling, extracorporeal shock wave therapy (ESWT), intense therapeutic ultrasound). Operative treatment is indicated when pain and functional limitations persist despite an adequate nonoperative trial lasting at least 6 months (Partial Plantar Fasciotomy-Gastrocnemius Lengthening) Radiofrequency (RF) that aims to reduce pain by targeting nerves . There are two main types: thermal RF ablation, which uses heat to damage nerve endings, and pulsed RF ablation, which uses less heat to desensitize nerves with a lower risk of complications. radiofrequency ablation (RFA) has emerged as a minimally invasive technique for the treatment of recalcitrant plantar fasciitis. RFA aims to disrupt pain transmission by targeting nerve tissue . There are two types of RFA: thermal radiofrequency ablation (TRFA) and pulse radiofrequency ablation (PRFA). TRFA involves the use of high temperatures to desensitize nerve endings, aiming to reduce pain by disrupting pain 4 signal transmission. However, the use of high temperatures carries a risk of damaging surrounding tissues, potentially leading to side effects and complications . PRFA, on the other hand, utilizes low-temperature pulsed electric fields to achieve nerve ablation in a less invasive manner. PRFA's neurodestructive effects are minimal, reducing pain without damaging surrounding soft tissues. The relatively long pauses between pulses in PRFA prevent excessive heating of nerve tissue, thus providing pain management without causing nerve damage. Compared to thermal RFA, PRFA has a minimal risk of causing neuritis, neuroma, and deafferentation pain(6) Steroids is a corticosteroid with potent anti-inflammatory and analgesic properties.

It has been shown to prolong the duration of sensory block and reduce postoperative nausea and vomiting (7)

ELIGIBILITY:
Inclusion Criteria:

* 1.Adult patients aged 18-65 years 2.ASA Physical Status I-II 3. patients diagnosed with chronic plantar fascitis

Exclusion Criteria:

* 1.patient refusal 2.Allergy to any study drug 3.pregnant , lactating women 4.Having undergone a prior surgery in the heel area/region 5.Having a history of trauma or fracture of the calcaneus 6.Having peripheral vascular ischemia 7.Having peripheral neuropathy and radiculopathy proven by electromyography or physical examination 8.Having calcaneal lesions, including benign tumors 9.Having an open wound or infection in the heel area/region 10.Having severe fat pad atrophy, calcaneal bursitis, and skin abnormalities around the heel 11.Having severe arthritic changes 12. bleeding disorder or on anti coagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
severity of pain | 24 hours after intervention
  NRS score can refer to a Numerical Rating Scale for pain , using a scale of 0-10 to measure severity, 0: No pain ,1-3: Mild , 4-6: Moderate and 7-10: Severe